CLINICAL TRIAL: NCT06864793
Title: A Randomized, Double-blind, Two-Period, Crossover Study to Compare the Pharmacokinetics and Safety of Recombinant Human Follicle Stimulating Hormone Injection (QL1012D) and Gonal-F® in Healthy Female Volunteers
Brief Title: Study on the Pharmacokinetics and Safety of QL1012D and Gonal-F® in Healthy Female Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: QL1012D-101
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A QL1012D (Experimental)
  Interventions: Drug: QL1012D
- Arm B Gonal-F® (Active Comparator)
  Interventions: Drug: Gonal-F®

INTERVENTIONS:
Drug: QL1012D — A single Subcutaneous injection, 225IU
  Other Names: Follitropin alfa
  Arms: Arm A QL1012D
Drug: Gonal-F® — A single Subcutaneous injection, 225IU
  Other Names: Follitropin alfa
  Arms: Arm B Gonal-F®

SUMMARY:
The goal of this Interventional study is to Compare the Pharmacokinetics and Safety of Recombinant Human Follicle Stimulating Hormone Injection (QL1012D) and Gonal-F® in Healthy Female Volunteers. It aims to evaluate the bioequivalence of recombinant human follicle stimulating hormone injection (QL1012D) and Gonal-F®, both given subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Female, Age between 18 to 45 years (inclusive).
* Body mass index (BMI) of ≥18 and ≤28 kg/m2, body weight ≥45 kg.
* With a history of sexual activity
* Regular menstruation cycle (25 to 35 days, inclusive).
* Normal sex hormone levels, or abnormalities deemed clinically insignificant by the investigator.
* Reached the standard within the time window after receiving the down-regulated drug.
* Agreed to take effective contraceptive measures during and 6 months after the end of the study period.
* Willing to participate in this clinical trial, understanding the study procedures, and able to provide written informed consent.

Exclusion Criteria:

* History of ovarian hyperstimulation syndrome, or polycystic ovary syndrome, or ovarian enlargement or cysts not caused by polycystic ovary syndrome, or primary ovarian failure; history of hypothalamic or pituitary tumors; history of malignancy; History of thrombosis; or other diseases that considered to influence the study by the investigator.
* Unexplained reproductive tract bleeding.
* Thin-layer cytology examination deemed clinically significant by the investigator.
* Vital signs, physical examination, 12-lead electrocardiogram, or laboratory examination deemed clinically significant by the investigator with.
* Pregnancy or lactation period, or positive human chorionic gonadotropin (HCG) examination.
* Known to be allergic to follicle-stimulating hormone (FSH), or gonadotropin-releasing hormone agonists (GnRH-a) or their analogs
* Consume strong coffee or tea daily
* Historic abuse of alcoholic beverages
* Smoke ≥5 cigarettes per day within 3 months prior to the study
* History of drug abuse
* Unsuitable for participation by the investigator.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cmax (maximum plasma concentration) | First Period: From pre-dose (0 hour) to 216 hours post-dose on Day 1. Second Period: From pre-dose (0 hour) to 216 hours post-dose on Day 11
  Maxmum observed serum concentration (Cmax) of QL1012D＆Gonal-f® in healthy Chinese female subjects.
AUC (area under the curve) | First Period: From pre-dose (0 hour) to 216 hours post-dose on Day 1. Second Period: From pre-dose (0 hour) to 216 hours post-dose on Day 11
  Adjusted geometric means of area under the serum concentration-time curve (AUC) of QL1012D＆Gonal-f® in healthy Chinese female subjects.